CLINICAL TRIAL: NCT05954871
Title: A Phase Ib Study to Evaluate the Safety, Pharmacokinetics, and Activity of GDC-1971 in Combination With Either Osimertinib in Patients With Unresectable, Locally Advanced, or Metastatic Non-Small Cell Lung Cancer, or With Cetuximab in Patients With Metastatic Colorectal Cancer
Brief Title: Study to Evaluate the Safety, Pharmacokinetics, and Activity of GDC-1971 in Combination With Either Osimertinib in Participants With Unresectable, Locally Advanced, or Metastatic Non-Small Cell Lung Cancer, or With Cetuximab in Participants With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO44272; 2022-502530-10-00 (Other: EU Clinical Trial Number)
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose-Finding Stage: Non-Small Cell Lung Cancer (NSCLC) (Experimental): Participants with unresectable, locally advanced or metastatic NSCLC will receive GDC-1971 at an assigned dose, orally, once daily (QD), on Days 1 to 28 of each 28-day cycle in combination with osimertinib, 80 milligrams (mg), orally, QD, on Days 1 to 28 of each cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: GDC-1971; Drug: Osimertinib
- Dose-Finding Stage: Colorectal Cancer (CRC) (Experimental): Participants with metastatic CRC will receive GDC-1971, at an assigned dose, orally, QD, on Days 1 to 28 days of each 28-day cycle in combination with cetuximab, 500 milligrams per square meter (mg/m^2), given by IV infusion on Days 1 and 15 of each cycle, until disease progression or unacceptable toxicity.
  Interventions: Drug: GDC-1971; Drug: Cetuximab
- Dose Expansion Stage: NSCLC (Experimental): Participants with unresectable, locally advanced or metastatic NSCLC will receive GDC-1971 at a dose determined in the dose finding stage, orally, QD, on Days 1 to 28 of each 28-day cycle in combination with osimertinib, 80 mg, orally, QD, on Days 1 to 28 of each cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: GDC-1971; Drug: Osimertinib
- Dose Expansion Stage: CRC (Experimental): Participants with metastatic CRC will receive GDC-1971 at a dose determined in the dose finding stage, orally, QD, on Days 1 to 28 of each 28-day cycle in combination with cetuximab, 500 mg/m^2, given by IV infusion on Days 1 and 15 of each cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: GDC-1971; Drug: Cetuximab

INTERVENTIONS:
Drug: GDC-1971 — GDC-1971 capsules or tablets will be administered as specified in each treatment arm.
  Other Names: RO7517834, RLY-1971
Drug: Osimertinib — Osimertinib tablets will be administered as specified in each treatment arm.
  Arms: Dose Expansion Stage: NSCLC; Dose-Finding Stage: Non-Small Cell Lung Cancer (NSCLC)
Drug: Cetuximab — Cetuximab, solution for infusion will be administered as specified in each treatment arm.
  Arms: Dose Expansion Stage: CRC; Dose-Finding Stage: Colorectal Cancer (CRC)

SUMMARY:
The main purpose of the study is to evaluate the safety of GDC-1971 in combination with either osimertinib or cetuximab. The study consists of a dose-finding stage followed by an expansion stage.

ELIGIBILITY:
Inclusion Criteria:

* Evaluable or measurable disease per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of ≥12 weeks
* Adequate hematologic and organ function within 14 days prior to initiation of study Inclusion Criteria for Non-Small Cell Lung Cancer Cohorts
* Histologically confirmed unresectable, locally advanced or metastatic adenocarcinoma of the lung that has progressed on/after prior treatment with third-generation epidermal growth factor receptor (EGFR) inhibitor (e.g., osimertinib)
* Positive for an EGFR exon 19 deletion or exon 21 L858R mutation
* Negative for acquired on-target EGFR alterations Inclusion Criteria for Colorectal Cancer Cohorts
* Histologically confirmed metastatic adenocarcinoma of the colon or rectum that has progressed on/after prior treatment with an EGFR inhibitor (e.g., cetuximab or panitumumab)
* Negative for kirsten rat sarcoma viral oncogene homolog (KRAS) alterations
* Negative for neuroblastoma RAS viral oncogene homolog (NRAS) alterations
* Negative for proto-oncogene B-Raf (BRAF) V600E alterations
* In lieu of a fresh pre-treatment biopsy, a recently obtained biopsy performed after completion of osimertinib therapy will be acceptable

Exclusion Criteria:

* Treatment with chemotherapy, immunotherapy, biologic therapy, or an investigational agent as anti-cancer therapy within 3 weeks or 5 drug elimination half-lives, whichever is shorter, prior to initiation of study treatment
* Treatment with endocrine therapy within 2 weeks prior to initiation of study drug, except for hormonal therapy with gonadotropin-releasing hormone agonists or antagonists for endocrine-sensitive cancers
* Significant traumatic injury or major surgical procedure within 4 weeks prior to Cycle 1, Day 1
* Positive hepatitis C virus (HCV) antibody test at screening
* Positive hepatitis B surface antigen (HBsAg) test at screening
* Known HIV infection
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Uncontrolled hypercalcemia
* Substance abuse, as determined by the investigator, within 12 months prior to screening
* Poor peripheral venous access
* Inability or unwillingness to swallow pills
* Malabsorption syndrome or other condition that would interfere with enteral absorption Chronic diarrhea, short bowel syndrome, or significant upper GI surgery including gastric resection, a history of inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis), or any active bowel inflammation (including diverticulitis)
* Serious infection within 4 weeks prior to screening
* History of malignancy within 3 years prior to screening
* Known and untreated, or active central nervous system (CNS) metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control)
* Leptomeningeal disease or carcinomatous meningitis
* History or presence of an abnormal electrocardiogram (ECG) that is deemed clinically significant by the investigator (e.g., complete left bundle branch block, second- or third-degree atrioventricular heart block) or evidence of prior myocardial infarction
* Left ventricular ejection fraction (LVEF) less than the institutional lower limit of normal (LLN) or <50%
* History or evidence of ophthalmic disease
* History of or active clinically significant cardiovascular dysfunction
* History of pulmonary firbrosis, organizing pneumonia, or pneumonitis

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 | Up to approximately 41 months
Number of Participants with Dose-Limiting Toxicities (DLTs) | Day 1 through Day 28 of Cycle 1 (1cycle= 28 days)

SECONDARY OUTCOMES:
Plasma Concentration of GDC-1971 | Up to approximately 41 months
Plasma Concentration of Osimertinib | Up to approximately 41 months
Objective Response Rate (ORR) as Determined by Investigator According to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1). | Up to approximately 41 months
Duration of Response (DOR) as Determined by Investigator According to RECIST v1.1 | Up to approximately 41 months
Progression-Free Survival (PFS) After Enrollment as Determined by Investigator According to RECIST v1.1 | Up to approximately 41 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- United States (2):
  - SCRI Oncology Partners, Nashville, Tennessee
  - START South Texas Accelerated Research Therapeutics-San Antonio, San Antonio, Texas
- Australia (2):
  - Border Medical Oncology, Wodonga, New South Wales
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).